CLINICAL TRIAL: NCT06752265
Title: Sexual Abuse Prevention Application On Children And Adolescents (Application Of Peran Sadar) Based On Empowering Parents And School Teachers In West Java
Brief Title: Application for Sexual Abuse Prevention Based On Empowerment of Parents And School Teachers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NURS-202406.01
Record Dates: First submitted 2024-11-17; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Child Abuse; Parents; Teachers
Keywords: Children; Application; Sexual abuse; Prevention; Adolescents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- child sexual abuse (Experimental): This group is an intervention group that will be given the PERAN SADAR intervention
  Interventions: Behavioral: Peran sadar application

INTERVENTIONS:
Behavioral: Peran sadar application — The PERAN SADAR application is an android-based SACA prevention application containing material related to SACA prevention which is given in a series for nine days using multimedia video stories and songs, documents, and tiktok in an attractive package, so that it attracts someone's interest in listening to the contents of the message. Social media applications are educational methods that are popular with all ages

SUMMARY:
The objective of the research is to Analyze the influence of providing the PERAN SADAR Application on the knowledge, attitudes, self-awareness, and communication practices of parents, teachers, children, and adolescents

Participants will get education that is given using the PERAN SADAR_ APPLICATION for 9 consecutive days. Teachers at school and parents at home were encouraged to provide information on preventing sexual abuse to their children after they had read and listened to the information in the PERAN SADAR_ Application. Information was given every day for 1 month. Children were given a knowledge questionnaire (which had been tested for validity and construct in previous studies) before being given an intervention to provide information on preventing sexual violence. After 1 month, knowledge, attitudes, self-awareness, and communication practices were measured for teachers and parents, while knowledge measurements were carried out for children.

ELIGIBILITY:
Inclusion Criteria:

* student at elementary school

Exclusion Criteria:

* sick, refuse to join

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 88 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge | one month
  Knowledge is the knowledge that parents and teachers have about sexual abuse. The Knowledge Questionnaire used is the Child Sexual abuse Prevention questionnaire for parents and teachers. This questionnaire consists of 30 multiple choice questions, given to parents and teachers before and after the intervention.
Attitudes | one month
  Attitudes towards preventing sexual abuse are views, feelings, and actions that reflect responsibility, and commitment to avoid, reduce, and stop all forms of sexual violence. The Attitude Questionnaire used is the Child Sexual abuse Prevention questionnaire for parents and school teachers. This questionnaire consists of 13 questions ranging from strongly agree to strongly disagree, this questionnaire was also given before and after the intervention
Self-Awareness | one month
  Self-awareness in the context of preventing sexual abuse is a person's ability to recognize, understand, and manage their own feelings, personal boundaries, and actions in order to protect themselves from risky or threatening situations, while preventing themselves from becoming perpetrators or causes of sexual abuse. The Self-Awareness Questionnaire used is the Self-Awareness Questionnaire for Preventing Sexual abuse in Children for Parents and School Teachers. This questionnaire consists of 20 questions ranging from strongly agree to strongly disagree, this questionnaire is also given before and after the intervention
Communication practices | one month
  Communication practice in preventing sexual abuse by parents and teachers to children is a systematic effort to build open, effective, and empathetic communication patterns with children, in order to provide education, understanding, and support needed to prevent sexual violence. The questionnaire used is the Communication Practices for Preventing Sexual abuse in Children questionnaire for parents and school teachers. This questionnaire consists of 17 multiple choice questions, this questionnaire was also given before and after the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Classroom, Sumedang, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Solehati T, Hermayanti Y, Bin Hazmi H, Trisyani M, Yusuf M, Kosasih CE, Nurfirdausi Islamah R. Empowering Children Through a Mobile Application for Sexual Abuse Prevention: The Supporting Roles of Parents and Teachers in a Cluster-Randomized Controlled Trial in Indonesia. J Multidiscip Healthc. 2025 Oct 3;18:6343-6360. doi: 10.2147/JMDH.S530036. eCollection 2025. PMID 41064336